CLINICAL TRIAL: NCT04929808
Title: Evaluation of a Novel Skin Care Product for the Management of Acute Radiodermatitis in Breast Cancer Patients
Brief Title: Novel Skin Care Product for the Management of Acute Radiodermatitis
Acronym: RTSkin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Collaborators: Hasselt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/058
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Radiodermatitis; Acute; Radiation Dermatitis
Keywords: Skin toxicity; Radiotherapy; Oncology; Skin care; Emollient
MeSH Terms: conditions — Radiodermatitis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Will receive the standard institutional skin care for acute radiodermatitis
  Interventions: Other: Standard institutional skin care
- Experimental group (Experimental): Will receive the novel, self-prepared skin care product
  Interventions: Other: Hydrating emollient for acute radiodermatitis

INTERVENTIONS:
Other: Hydrating emollient for acute radiodermatitis — The emollient has a calming effect, and hydrating and anti-oxidative properties.
  An absorbable wound dressing will be applied on painful and moist wounds. In case of severe itch, a systemic antihistaminic agent can be prescribed by the radiotherapist.
  Arms: Experimental group
Other: Standard institutional skin care — The control patients will receive the institutional standard skin care, which includes the application of Flamigel® (Flen Pharma, Kontich, BELGIUM). In addition, Mepilex® (Mölnlycke Health Care, Berchem, Belgium), an absorbable wound dressing will be applied on painful and moist wounds. In case of severe itch, a systemic antihistaminic agent can be prescribed by the radiotherapist.
  Arms: Control group

SUMMARY:
Notwithstanding the continuous progress in cancer treatment, patients with cancer still have to cope with quality of life (QoL) - impairing complications. Especially an extensive spectrum of dermatologic toxicities has been associated with cancer treatments. The number and type of cutaneous toxicities have evolved over the past 50 years, paralleling the development of new radiotherapy (RT) techniques. Acute radiodermatitis (ARD) is a distressing and painful skin reaction that occurs in 95% of the patients undergoing RT.

Important organizations in the field of oncology and supportive care, such as the MASCC, the ASCO, and the ESMO, have developed guidelines for the management of cancer therapy- related cutaneous toxicities based on available scientific evidence. Still, for some interventions, the evidence of recommendation is moderate to insufficient. Therefore, it is essential to elucidate other new potential management strategies for dermatological complications of cancer treatment. Based on the previously mentioned supportive care guidelines for the RTskin project, a novel emollient to tackle ARD has been developed.

The RTskin project general aim is to evaluate the efficacy of a novel skincare product to manage ARD in breast cancer patients.

DETAILED DESCRIPTION:
Primary objective Evaluate the efficacy of a novel emollient for the management of ARD in comparison with the current standard of care in breast cancer patients

Secondary Objective 1 Compare the ARD-related symptoms of in breast cancer patients treated with the novel emollient and the standard institutional skin care.

Secondary Objective 2 Compare the dermatologic quality of life of in breast cancer patients treated with the novel emollient and the standard institutional skin care.

Secondary Objective 3 Correlate the severity of ARD with the applied RT parameters and personal - medical characteristics

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer and underwent lumpectomy or mastectomy
* Scheduled for radiotherapy: hypofractionation regimen (16 or 16+5 boost fractions) at the Jessa Hospital (Hasselt, BE)
* Age ≥ 18 years
* Able to comply to the study protocol
* Able to sign written informed consent
* Signed written informed consent

Exclusion Criteria:

* Previous irradiation to the breast region
* Metastatic disease
* Patients with pre-existing skin rash, ulceration or open wound in the treatment area
* Substance abuse patients or patients with medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results as judged by the investigator •- Any condition that is unstable or could affect the safety of the patient and their compliance in the study as judged by the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Skin reaction evaluation | Baseline
  The patients skin reactions will be evaluated by the modified version of the RTOG criteria
Skin reaction evaluation | At fraction 15-16 of radiotherapy (week 3 )
  The patients skin reactions will be evaluated by the modified version of the RTOG criteria
Skin reaction evaluation | At fraction 20-21 of radiotherapy (week 4) in case of a tumor boost
  The patients skin reactions will be evaluated by the modified version of the RTOG criteria

SECONDARY OUTCOMES:
Patient subjective evaluation of skin reactions | Baseline
  The patients will be asked to complete a questionnaire to evaluate the intensity and frequency of five common symptoms of skin reactions: pruritus, dryness, erythema, burning sensation, and pain on an 11-point Numerical Rating Scale
Patient subjective evaluation of skin reactions | Week 1 of radiotherapy
  The patients will be asked to complete a questionnaire to evaluate the intensity and frequency of five common symptoms of skin reactions: pruritus, dryness, erythema, burning sensation, and pain on an 11-point Numerical Rating Scale
Patient subjective evaluation of skin reactions | Week 2 of radiotherapy
  The patients will be asked to complete a questionnaire to evaluate the intensity and frequency of five common symptoms of skin reactions: pruritus, dryness, erythema, burning sensation, and pain on an 11-point Numerical Rating Scale
Patient subjective evaluation of skin reactions | At fraction 15/16 of radiotherapy (week 3)
  The patients will be asked to complete a questionnaire to evaluate the intensity and frequency of five common symptoms of skin reactions: pruritus, dryness, erythema, burning sensation, and pain on an 11-point Numerical Rating Scale
Patient subjective evaluation of skin reactions | At fraction 20/21 of radiotherapy (week 4) in case of a tumor boost
  The patients will be asked to complete a questionnaire to evaluate the intensity and frequency of five common symptoms of skin reactions: pruritus, dryness, erythema, burning sensation, and pain on an 11-point Numerical Rating Scale
Quality of life assessment | Baseline
  The skindex-29 is a validated instrument to measures patients' QoL specifically correlated with skin conditions. It has 3 scales addressing emotions (10 items), symptoms (7 items) and functioning (12 items).
Quality of life assessment | At fraction 15/16 of radiotherapy (week 3)
  The skindex-29 is a validated instrument to measures patients' QoL specifically correlated with skin conditions. It has 3 scales addressing emotions (10 items), symptoms (7 items) and functioning (12 items).
Quality of life assessment | At fraction 20/21 of radiotherapy (week 4) in case of a tumor boost
  The skindex-29 is a validated instrument to measures patients' QoL specifically correlated with skin conditions. It has 3 scales addressing emotions (10 items), symptoms (7 items) and functioning (12 items).
Patients' satisfaction with the therapeutic intervention | At fraction 15/16 of radiotherapy (week 3)
  The patients will be asked to evaluate the general pleasantness and soothing effect of the skin care products. Furthermore, they will be asked to score their global satisfaction with the skin care products. All these items will be evaluated by using a numerical rating scale (NRS).
Patients' satisfaction with the therapeutic intervention | At fraction 20/21 of radiotherapy (week 4) in case of a tumor boost
  The patients will be asked to evaluate the general pleasantness and soothing effect of the skin care products. Furthermore, they will be asked to score their global satisfaction with the skin care products. All these items will be evaluated by using a numerical rating scale (NRS).
Pruritus evaluation | Baseline
  The patients' degree of pruritus will be evaluated by the NCI-CTCAE V5 criteria
Pruritus evaluation | At fraction 15/16 of radiotherapy (week 3)
  The patients' degree of pruritus will be evaluated by the NCI-CTCAE V5 criteria
Pruritus evaluation | At fraction 20/21 of radiotherapy (week 4) in case of a tumor boost
  The patients' degree of pruritus will be evaluated by the NCI-CTCAE V5 criteria

OTHER OUTCOMES:
General patient-, disease-, and treatment-related information | Baseline
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (i.e., gender, age, smoking history, work habits, physical activity, skin condition, alcohol use, and medication use). Furthermore, information about disease- and treatment-related risk factors will be collected through medical records (e.g., tumor type and stage, tumor site, treatment type, radiotherapy regime.
General patient-, disease-, and treatment-related information | Week 4 of radiotherapy
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (i.e., gender, age, smoking history, work habits, physical activity, skin condition, alcohol use, and medication use). Furthermore, information about disease- and treatment-related risk factors will be collected through medical records (e.g., tumor type and stage, tumor site, treatment type, radiotherapy regime.
General patient-, disease-, and treatment-related information | Two weeks post-radiotherapy (follow-up)
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (i.e., gender, age, smoking history, work habits, physical activity, skin condition, alcohol use, and medication use). Furthermore, information about disease- and treatment-related risk factors will be collected through medical records (e.g., tumor type and stage, tumor site, treatment type, radiotherapy regime.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Mebis, MD, PhD, Principal Investigator — Jessa ziekenhuis VZW
Locations (1):
- Jessa Ziekenhuis VZW, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robijns J, Van Bever L, Hermans S, Claes M, Lodewijckx J, Lenaerts M, Tuts L, Vandaele E, Vinken E, Noe L, Verboven K, Maes A, Van de Velde AS, Bulens P, Bulens P, Van den Bergh L, Mebis J. A novel, multi-active emollient for the prevention of acute radiation dermatitis in breast cancer patients: a randomized clinical trial. Support Care Cancer. 2023 Oct 11;31(12):625. doi: 10.1007/s00520-023-08096-5. PMID 37819539